CLINICAL TRIAL: NCT04411355
Title: Nursing Management in Patients With Hypertension
Brief Title: The Effect of Chronic Care Model Based Education on Disease Management in Hypertensive Patients
Acronym: CCM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gülbin Konakçı, Asst. Prof., Ege University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 494582
Record Dates: First submitted 2020-05-11; First posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Hypertension
Keywords: nursing; chronic care model; hypertension
MeSH Terms: conditions — Hypertension | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: controlled semi-experimental design in matched groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group patients (No Intervention): non intervention. only rutin care
- intervention group patients (Experimental): The intervention group was trained and monitored by a professional team in line with the components of the model. Life quality scale, hypertension information questions and chronic care assessment scale were applied to both groups at the beginning and in the sixth month of the study.
  Interventions: Dietary Supplement: control by dietitian; Other: Exercise programs; Behavioral: control by psychiatrist

INTERVENTIONS:
Dietary Supplement: control by dietitian
  Other Names: behavioral
  Arms: intervention group patients
Other: Exercise programs — In line with the address information of the intervention patients, purpose/content of the study was discussed with the gyms of municipalities and patients were made to benefit from these facilities for free. For the patients preferring private gyms, it was ensured that discounts were made for the patients.
  Arms: intervention group patients
Behavioral: control by psychiatrist — The psychiatrist assessed the suitability of the patients to the study, assessed the patients having adaptation problems with respect to lifestyle changes in monthly controls and also played roles in teaching the coping methods to patients and applying and interpreting the hospital anxiety and depression scale.
  Arms: intervention group patients

SUMMARY:
Background: This study was conducted to examine the effect of planned educational intervention based on The Chronic Care Model (CCM) on the management of hypertension in patients with hypertension. The Chronic Care Model is a framework for organizing and improving chronic illness care, based on a proactive, planned approach that incorporates patient self-care, provider, and system level interventions. Several instruments have been developed to evaluate the effects of CCM implementation on care and treatment outcomes.The Patient Assessment of Chronic Illness Care (PACIC) questionnaire is used in instrument to evalate the delivery of care for patients.

Methods: The study was performed a prospective and conducted with a controlled semi-experimental pattern in matched groups. 30 patients including 15 intervention and 15 control group patients matched in terms of socio-demographic features were monitored for six months. The intervention group was trained and monitored by a professional team in line with the components of the model. Life quality scale, hypertension information questions and chronic care assessment scale were applied to both groups at the beginning and in the sixth month of the study.

Trial registration: The study was conducted in accordance with the World Medical Association Declaration of Helsinki of 1964, and approved by local authorities and local Bioethics Committees(BC) in participating university hospital. (Ethics committee approval No:B.30.2.EGE.0.20.05.00/OY/649/268 Decision No: 13-3.3/12) Permissions for the use of scale of PACIC and model of CCM were taken via e-mail.

Key Words: nursing; chronic care model; hypertension

DETAILED DESCRIPTION:
According to the World Health Organisation, 60% of all deaths in the world result from chronic illnesses, and 80% of these deaths occur in low and middle income countries (WHO 2008a).One of the most common chronic illnesses is hypertension, and it affects almost 20% of the adult population. The fact that chronic diseases have become widespread nowadays reveals the importance of chronic disease control and community-based disease management programs (Cranston 2006). Chronic disease management includes the treatment of the disease and preparing and strengthening the patients to help patients to gain self-management skills. With an effective disease management; symptoms, recourses to emergency units and hospitalisation can be reduced, physiological and psychological effects of the disease can be limited, dependence can be prevented, and life quality can be enhanced (Haskett 2006). Among the models of chronic disease management, the most well-known, the most frequently used and the most effective one is "Chronic Care Model"(CCM) (Piat et al. 2007). Since social and economic burden has gradually increased in chronic care management, "CCM" was presented as a guide with the aim of enhancing the quality of the care and reducing the care costs (Geyman 2007). The main point of the model identified by Wagner et al. is the "existence of a fruitful interaction between the health care team and the patient" (Rothman & Wagner 2003, Solberg et al. 2005). According to the model, the "patient" motivated by a relation of knowledge, skill and trust and the "health care team" having the necessary expertise, knowledge and sources can take effective decisions for a high quality care and conduct an effective chronic disease care management by using the available sources (ICN 2010, Wagner 2001). This research was conducted to evaluate the effects of the use of the CCM in patients with hypertension on life quality and clinic results and to conduct a study concerning the use of this model in the chronic diseases in Turkey.

METHODS Research Design:The research was conducted in the nephrology polyclinic of a university hospital for six months with a controlled semi-experimental design in matched groups.

Population and sample:Population of the research consisted of all patients who applied to and followed in the nephrology polyclinic. In the selection of the sample, patient files were listed by using the polyclinic records. Out of this list,2 groups were created as intervention and control group matched in consideration of socio-economic variables such as age, sex and educational background. According to the power-analysis method, 15 intervention and 15 control group patients constituted the sample of the research. The power of the study was determined as 90% in p=0,05 reliability coefficient .

Data collection tools:In collecting the data, researcher used the socio-demographic features form prepared in consideration of the literature and expert views and the following forms for follow-up.

Attitude and habits scale concerning hypertension Information about hypertension WHOQOL-BREF(Tr) life quality assessment scale Chronic Disease Care Assessment Scale (PACIC) Hospital Anxiety and Depression Scale Integration of CCM into the study I. Organization of Health Care

1. Multidisciplinary Team and Duties and Responsibilities Multidisciplinary team consisted of internal medicine specialist, internal medicine specialist nurse, dietician and psychologist. Consultation was required from the other areas of specialisation when needed.

   Team Members (Primary Care Team): Internal medicine specialist carried out the physical examinations and system diagnosis of the patients to be included in the study, determined the laboratory requests and assessed the monthly patient data and shared the results with the team. The internal medicine specialist nurse collected and assessed the data, planned and executed the training, arranged weekly interviews and monthly controls and assessed the data. The psychiatrist assessed the suitability of the patients to the study, assessed the patients having adaptation problems with respect to lifestyle changes in monthly controls and also played roles in teaching the coping methods to patients and applying and interpreting the hospital anxiety and depression scale. Dietician planned the diet programs together with the patients and determined the calorie needs of diet programs.
2. Identification of Objectives and Expected Results:

The objectives of this study were determined in line with the following points that are considered to have impact on the success of the disease management:

i.Since hypertension is a chronic disease, its management requires a long and effective time.

ii.In the management of hypertension, patient is prioritised, not the disease. It requires a multidisciplinary teamwork with the patient, and team members need to work in an effective and cooperative manner.

iii.It is important to determine the lifestyle and habits ofthe patient in the treatment of hypertension. Each patient diagnosed with hypertension display different behaviours and thus, different approaches might be needed for each patient.

iv.Care and follow-up plans should be developed by determining the compliance/incompliance of patients to treatment and lifestyle changes, and the trust of the patient to care and treatment team is important in compliance to disease.

v.Health education should be constant and accessible in hypertension; behavioural change takes time and therefore, it requires follow-up and motivation.

vi.Patient education is planned in consideration of the faith and cultural values of the patient.

c.Metabolic Control Variables were determined as fasting plasma glucose, serum total cholesterol, Serum LDL-cholesterol, Serum HDL- cholesterol, fasting serum triglycerides, HbA1C, spot urine, Glomerular filtration rate, ECG, height, weight, waist circumference and BMI.

At the end of the study where the above mentioned points were addressed, it was expected that the patients could implement the lifestyle changes, could be effective in disease management, improvements would be observed in metabolic indicators related to the disease, adaptation of patients to disease and treatment and patients' life qualities would be improved, and patients' perspectives to the healthcare team would change.

II.Self-management support: A training manual was prepared for information about the disease while PowerPoint presentations were prepared for individual trainings. Data collection forms were applied to determine the factors affecting compliance with the treatment, and data were shared with the patients.

Training manual, PowerPoint presentation and web education page Socio-Demographic Features Data Form Metabolic values form Form for assessing the attitude and habits related to hypertension Information about hypertension WHOQOL-BREF(Tr) quality of life assessment form Patient Assessment of Chronic Illness Care (PACIC) Hospital Anxiety and Depression Scale III.Delivery System Design In both control and intervention groups, data forms were filled out at the beginning (0th month) and at the end (6. month) of the study. An intermediate control was carried out in the 3rd month for metabolic values. For the patients in the intervention group, trainings planned for lifestyle changes and disease management were delivered. No training was provided to the control group.However, at the end of the study, all trainings and information were provided to the patients in the control group.During preparation, a web page was designed to start the web-based training to the patients in the intervention group through internet connection from intervention group houses. In the hospital where the study was conducted, a database which could be accessed only with a personal password and the team members followed the patients through this database.Tension measuring training was provided to the patients in the intervention group by using 5A method so that the follow-up form could be used at home.

Through phone calls, patients were encouraged to comply with the program. Situations preventing the compliance of patients and solution proposals were discussed. Activities which will enable participants to use their social supports effectively were discussed, as well. Calls were made by the researcher in charge and recorded in the patient database IV. Decision Support: Evidence-based manuals were used in the patient and patient relative training. Turkish Society of Cardiology National Hypertension Treatment and Follow-up Manual (2000), Turkish Society of Cardiology Nursing Care Manual for Heart Failure, Acute Coronary Syndromes and Hypertension (2007), European Society of Cardiology (ESC) Arterial Hypertension Treatment Manual 2007, Pulmonary Hypertension Diagnosis and Treatment Manual (2009), ACC/AHA Hypertension in the Aged Manual (2011), WHO-ISH (World Health Organisation/International Society for Hypertension 2003 Manual, JNC-7 2003 (Joint Committee 7th Report- USA Hypertension Manual), Turkish Society of Hypertension and Renal Diseases, Hipder TRNC Hypertension Society, webpage of the Ministry of Health Public Health Institution of Turkey,Information manual, Web-based training (www.ygulbin.com).

V.Clinical Information Systems: An electronic patient file was created for each patient included in the study in the database taken from the data processing centre of the hospital (In this e-file, demographic characteristics of the patient, data collection tools used in the study and the data results, cardiovascular risk table, appointment dates, phone call results, patient assessment section reserved for each team member, consultation results, urgent and immediate intervention situations emerging during the study, comorbidity record are included). The database explained above can be accessed only through a password so that only team members can have access to data, interference in the study data is prevented, and patient privacy and confidentiality are protected as the ethical dimension of the study.

VI.Social resources and policies: Exercise programs: In line with the address information of the intervention patients, purpose/content of the study was discussed with the gyms of municipalities and patients were made to benefit from these facilities for free. For the patients preferring private gyms, it was ensured that discounts were made for the patients.

Statistical Analysis In the statistical analysis of the data, number and percentage distribution, significance test of the difference between two pairs (t test), significance test of the difference between two means (t test), one way variance analysis (ANOVA), chi-square test and Mann-Whitney U test, General Linear Model - repeated measures define Factor(s) at repeated measurements were used through Statistical Package for Social Sciences for Windows Version 18.0 software. Statistical analyses were carried out by a biostatistics expert.

Ethical Consents:Written and verbal consents were received from the patients for conducting the research.Ethics committee approval No:B.30.2.EGE.0.20.05.00/OY/649/268 Decision No: 13-3.3/12) was received from the institution where the study was conducted. Permissions for the use of scales and model were taken via e-mail. As ethical responsibility, the same training, training materials and exercise opportunities were provided to the patients in the control group at the end of the research. Since blood and urine tests and other examinations to be used in the study were performed in the polyclinics where patients received service during their routine controls, the patient or researcher was not charged a fee.

ELIGIBILITY:
Inclusion Criteria:* Being in the 18-65 age group

* Being literate
* No sensory losses such as vision and hearing
* Willingness to participate in the study
* Being open to communication and cooperation
* Internet access and availability
* To have a phone that can be reached
* Having a diagnosis of hypertension at least 6 months ago
* According to JNC-6,1997 classification, high blood pressure level is normal, stage 1,2 and 3, risk group A and B, no additional organ damage
* Not having metabolic disturbances or diseases that prevent to from participating in the study.

Exclusion Criteria:Not being a volunteer

* Not complying with inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-12-15 (Actual); Primary Completion 2014-02-15 (Actual); Study Completion 2016-04-15 (Actual)

PRIMARY OUTCOMES:
The Patient Assessment of Chronic Illness Care (PACIC) | 6 months
  The tool was developed in 2005 by Glasgow and is allowing the evaluation of health care services offered to chronic patients by patients,easy to apply,20 items short tool.PACIC,created in line with the basic 6 elements of the CCM,consists of 5 subdimensions;*Patient Activation (items 1-3),*Delivery System Design/Decision Support (items 4-6),*Goal Setting (items 7-11),*Problem-solving/Contextual Counseling (items 12-15),*Follow-up/Coordination (items 16-20).The total score of the scale is calculated by the average score of all 20 items.The average score of each sub-dimension are measured by a 5-point Likert-type grading. The increase in scale scores indicates that individuals with chronic diseases have high satisfaction with the care patients receive and that chronic disease management is sufficient.The validity and reliability of theTurkish version of the scale was done by İncirkuş and Nahcivan(2010).
WHOQOL-BREF(TR) quality of life assessment | 6 months
  The WHOQOL-BREF(TR)scale developed from WHOQOL-100 to evaluate the quality of life.The cultural adaptation of the scale inTurkey performed by Eser(1999).The Turkish versionof the scale,27th question,national environmental area has been added as"Area V"; Area I:Physical area:To be able to carry out daily tasks,dependence on drugs, treatment, vitality,fatigue,physical activity,pain,discomfortsleep,rest,ability to work.
  Area II:Mental area:Body image and appearance,negative emotions,memory, distraction.
  Area III:Social relations area:Relations with other people,social support,sexual life.
  Area IV:Environmental area:Financial resources,physical security,accessibility to health services,home environment,opportunity to use rest,leisure time,physical environment, transportation.
  Area V:National environmental area:cultural area The total score is range from a min.of 27 to a max.of 135.
Hypertensive nephropathy | 6 months
  The reduced glomerular filtration rate (eGFR). GFR rate is calculated using a mathematical formula that compares a person's size, age, sex, and race to serum creatinine levels. A normal GFR 60 mL/min/1.73 m² .the lower the GFR number, the worse the kidney function.

SECONDARY OUTCOMES:
HbA1c levels as the clinical indicator | 3. and 6. month
  The HbA1c test evaluates the average amount of glucose in the blood in the last 3 months.
  Traditionally, in our country, HbA1c is expressed as a percentage. The normal HbA1c value is between 4 and 6 mg/dl.
Blood glucose levels as the clinical indicator | 6. month
  peripheral blood will be checked and at least 8 hours fasting blood sugar level 70-100 mg/dl
The indicator of perfusion to vital organs | 6. month
  The mean arterial pressure (MAP) MAP = 1/3 (systolic blood pressure - diastolic blood pressure) + diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Huseyin Töz, prof, Study Director — Deparment of Nephrology of Ege University Hospital; Asiye Durmaz Akyol, Study Director — Faculty of Nursing of Ege University

IPD SHARING:
Plan to Share IPD: Yes
In the hospital where the study was conducted, a database which could be accessed only with a personal password and the team members followed the patients through this database.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: open-ended
Access Criteria: unconditional
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp

REFERENCES:
- See also: National Thesis Center — https://tez.yok.gov.tr/UlusalTezMerkezi
- Available data/document: National Thesis Center: 10128359 — https://tez.yok.gov.tr/UlusalTezMerkezi — thesis Number: 494582